CLINICAL TRIAL: NCT00501462
Title: An Evaluation of the Pharmacokinetics of a Single Oral Dose of GSK189075 in Patients With Varying Degrees of Renal Insufficiency Compared to Volunteers With Normal Renal Function
Brief Title: A Comparison Of Study Drug Blood Levels After One Dose Of GSK189075 In Subjects With Normal And Reduced Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KG2105253
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-06

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 2; Renal Insufficiency
Keywords: Type 2 Diabetes Mellitus; renal insufficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mild renal impairmnent (Other)
  Interventions: Drug: GSK189075
- moderate renal impairment (Other)
  Interventions: Drug: GSK189075
- Normal renal function (Other)
  Interventions: Drug: GSK189075

INTERVENTIONS:
Drug: GSK189075 — single 250 mg dose of drug

SUMMARY:
This is an open-label study that will measure blood levels of different parts of a drug called GKS189075. People participating in this study will receive a single dose of 250mg GSK189075 by mouth. About 20 people with mild to moderate decrease in renal (kidney) function will be asked to participate in this study. They will be compared to about 20 healthy participants who are close to the same age and body size. People participating in this study will stay at a clinical research unit beginning 2 days before they receive their single dose of GSK189075 and will remain there until approximately one day after receiving the study drug. During this study urine will be collected beginning the day before receiving study drug until the day after, just prior to leaving the clinical research unit. Blood samples will also be collected at various times beginning immediately before until 24 hours after receiving the study drug.

ELIGIBILITY:
Inclusion Criteria:

* A female is eligible to enter and participate in this study if she is of Non-child-bearing potential with a negative pregnancy test at screening or of Childbearing potential, has a negative serum pregnancy test at screening, is not lactating, and agrees to adequate contraception.
* Satisfactory medical evaluation based upon medical history, medication history, physical examination, and clinical laboratory data obtained at the Screening visit.
* Body weight > 50 kg. BMI within the range of 19 to 40 kg/m2.
* Signed and dated written informed consent prior to participation in any protocol-specific procedures, including screening procedures.
* The subject is able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions.
* Additional Inclusion Criteria for Subjects with Renal Insufficiency: Subjects with renal insufficiency must be considered by the investigator to be clinically stable. Subjects must continue to meet this criterion of stable renal function upon check-in into the clinic

Exclusion Criteria:

* History of regular alcohol consumption averaging >7 drinks per week for women or >14 drinks per week for men within 6 months of Screening. One drink is equivalent to 12 g alcohol = 5 ounces (oz; 150 ml) of wine or 12 oz (360 ml) of beer or 1.5 oz (45 ml) of 80 proof distilled spirits.
* A positive drug or alcohol test at Screening or Check-in.
* Smokers will be allowed to enrol in the study; however, smoking that interferes with the collection/recording of ongoing study procedures will not be allowed. Smoking status will be recorded in the CRF.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication for the current study.
* The subject has donated more than 450mL blood within the 56 day period prior to the first scheduled administration of GSK189075.
* Known or suspected gastroparesis, gastric surgery within the 6 months prior to screening, or any other gastrointestinal condition that would likely interfere with absorption of GSK189075.
* Subjects with clinical laboratory values outside rages as specified in the protocols
* Any subject with either documented cirrhosis or a history consistent with a diagnosis of cirrhosis.
* Urinary tract or bladder infection within 4 weeks of the first scheduled administration of study drug.
* Positive hepatitis B surface antigen, or HIV at Screening. If negative test results have been documented within the last 2 months, it will not be necessary to repeat these tests. Subjects with positive results for hepatitis C antibodies may be eligible if they have normal liver enzymes and no history of hepatitis and are approved by the GSK medical monitor.
* Any history of myocardial infarction, cardiac syncope.
* A history of clinically significant cardiac arrhythmias (individual cases to be discussed with the GSK Medical Monitor).
* A history of unstable angina in the past 6 months.
* Cardiac conduction abnormalities denoted by ranges specified in the protocol
* Systolic blood pressure < 80 mmHg or > 180 mmHg
* Diastolic blood pressure < 60 mmHg or > 100 mmHg
* Use of prescription or non-prescription drugs (including high dose vitamins, herbal and dietary supplements [including St. John's Wort]) within 7 days prior to administration of the first dose of study medication, unless in the opinion of the investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety. Some allowable exceptions are found in the Permitted Medications section (Section 9.1).

Additional Exclusion Criteria for Subjects with Renal Insufficiency

* Patients on a new drug regimen (defined as starting a new drug or changing dosage regimen of a current drug within 7 days prior to administration of GSK189075). No restrictions will be placed on the use of insulin, 1,25 dihydroxyvitamin D3 (Rocaltrol), erythropoietin, and calcium- or aluminum-containing phosphate binders.
* Subjects whose current medication therapy is not in agreement with the information provided in Sections 9.1, 9.2, or 9.3 of this protocol.
* Serum albumin less than 2.5 g/dL.
* Hemoglobin less than 8.5 g/dL. Additional Exclusion Criteria for Subjects with Normal Renal Function
* Any clinically relevant abnormality identified on the screening physical or laboratory examination. Any abnormalities of outside the normal reference range at Screening may be repeated once and must be reviewed with the GSK Medical Monitor prior to enrollment of a subject into the study.
* Hemoglobin or hematocrit below the reference range at Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
drug & metabolite plasma levels | at 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, & 24 hours after dosing

SECONDARY OUTCOMES:
urine levels of Glucose & electrolytes, Drug & metabolites | at 0-6, 6-12 & 12-24 hours after dosing
ECG, labs, vital signs, adverse events | each visit
Plasma protein binding of GSK189074 and GSK279782 | 2 hr
GSK189074 and GSK279782 in 24 hour urine collection and corresponding renal clearance CLr. | 24 hr
urine glucose excreted. | 6, 12, 24 hours
Urinary creatinine clearance (CLcr). | 6, 12, 24 hours
Safety and tolerability parameters, including AEs and clinically relevant changes in vital signs (heart rate and blood pressure), ECGs, urine electrolytes, and clinical laboratory assessments (clinical chemistry, hematology, and urinalysis). | 1, 2, 4, 12, 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Austin, Texas